CLINICAL TRIAL: NCT06888986
Title: Integration of VR, AR, AI and Wearable Technology to Develop Innovative Health Education and Monitoring Systems on Symptom Management, Situational Reaction, Learinging Process and Physical and Psychological Health of Early Dementia
Brief Title: Integration of VR and AR Dementia Prevention Health Education Progrom for Older Adults With Mild Cognitive Impairment
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan Normal University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 202212HM033
Record Dates: First submitted 2025-03-11; First posted 2025-03-21 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Mild Cognitive Impairment (MCI); Dementia; Health Literacy; Self-Efficacy; Attitude to Health; Virtual Reality; Health Education; eHealth; Older Adults (65 Years and Older)
MeSH Terms: conditions — Cognitive Dysfunction; Dementia; Health Education

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (VR Dementia Prevention Education) (Experimental): Participants in this arm will take part in the VR Dementia Prevention Health Education Module, an immersive virtual reality (VR) intervention aimed at enhancing dementia-related knowledge, health literacy, self-efficacy, and attitudes toward dementia. The intervention combines 360-degree panoramic VR technology with interactive educational content to create a realistic and engaging learning experience for older adults with mild cognitive impairment (MCI).
  Interventions: Behavioral: VR Dementia Prevention Health Education Module
- Control Group (No Intervention) (No Intervention): Participants in this arm will not receive any active intervention during the study. They will continue with their usual daily routine, without exposure to VR-based health education or any structured dementia-related educational programs. This group serves as a comparison to evaluate the effects of the VR Dementia Prevention Health Education Module administered to the experimental group.

INTERVENTIONS:
Behavioral: VR Dementia Prevention Health Education Module — A virtual reality (VR) cognitive health education program designed to enhance knowledge related to dementia, improve health literacy, boost self-efficacy, and shape attitudes towards dementia. Participants engage with 360-degree immersive VR modules using VR headsets that simulate real-world scenarios related to dementia. The intervention comprises five interactive VR sessions, each addressing important topics in dementia prevention and management. Trained research staff will guide participants to ensure safe and effective interaction with the VR system.
  Arms: Experimental Group (VR Dementia Prevention Education)

SUMMARY:
The goal of this randomized controlled trial is to evaluate the effectiveness of Virtual Reality (VR)-based cognitive health education for older adults with mild cognitive impairment (MCI) in Taiwan. The study aims to assess whether VR-supported interventions improve cognitive health knowledge, health literacy, and self-management skills among participants.

The primary research questions are:

1. Does the VR-based intervention enhance participants' knowledge related to dementia and their health literacy?
2. Does the VR-based intervention improve cognitive function, mental well-being, and self-efficacy compared to a control group?

Participants will be randomly assigned to one of two groups:

1. Intervention group: This group will receive the "VR Dementia Prevention Health Education Module," an immersive virtual reality program designed to enhance dementia-related knowledge and coping strategies.
2. Control group: This group will receive standard, routine health education without VR exposure.

DETAILED DESCRIPTION:
This study is a randomized controlled trial (RCT) aimed at evaluating the effectiveness of a Virtual Reality (VR)-based cognitive health education program for older adults in Taiwan who show signs of mild cognitive impairment (MCI). The research seeks to determine whether VR-enhanced dementia prevention education increases dementia-related knowledge, health literacy, self-efficacy, and acceptance of dementia compared to a control group receiving standard health education without VR exposure and intervention.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 65 years and older.
* AD-8 score of 2 or higher, indicating possible cognitive impairment.
* Ability to understand and follow basic instructions in Mandarin or Taiwanese.
* Capacity to provide informed consent or have a legally authorized representative to provide consent.
* Ability to tolerate and interact with VR equipment (e.g., wearing a VR headset, using hand controllers).

Exclusion Criteria:

* Diagnosed with moderate to severe dementia (i.e., unable to follow basic instructions).
* Presence of severe visual, auditory, or motor impairments that hinder interaction with VR devices.
* Diagnosed with severe psychiatric disorders (e.g., schizophrenia, major depressive disorder).
* Unable to communicate effectively in Mandarin or Taiwanese.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-09-30 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in Dementia-Related Knowledge | Baseline (Day 0, prior to intervention start) Immediate Post-Intervention (Day 0, following completion of the VR session, approximately 2 hours after Baseline assessment) Follow-up (Month 3, 12 weeks post-intervention, to assess retention effects)
  Dementia-related knowledge will be assessed using the Dementia Knowledge Assessment Scale (DKAS), a validated tool for evaluating comprehensive understanding of dementia. The DKAS includes 25 true/false items and provides an additional "Don't Know" response option to reduce guessing.
Change in Health Literacy | Baseline (Day 0, prior to intervention start) Immediate Post-Intervention (Day 0, following completion of the VR session, approximately 2 hours after Baseline assessment) Follow-up (Month 3, 12 weeks post-intervention, to assess retention effects)
  Health literacy concerning dementia prevention will be evaluated using the Dementia Health Literacy Scale (DHLS). The DHLS includes 20 items rated on a 5-point Likert scale (1 = strongly disagree to 5 = strongly agree). This scale features three subdomains: Functional Health Literacy (8 items) - Evaluates the ability to manage dementia-related information for daily needs; Communicative Health Literacy (5 items) - Assesses skills in accessing, understanding, and applying dementia-related health information during interactions; and Critical Health Literacy (7 items) - Gauges higher-order cognitive skills and the ability to critically analyze dementia-related health information.

SECONDARY OUTCOMES:
Change in Self-Efficacy Related to Dementia Prevention | Baseline (Day 0, prior to intervention start) Immediate Post-Intervention (Day 0, following completion of the VR session, approximately 2 hours after Baseline assessment) Follow-up (Month 3, 12 weeks post-intervention, to assess retention effects)
  Self-efficacy will be assessed using the Dementia-Related Self-Efficacy Scale (DSES), which has been adapted from existing self-efficacy measures and validated through expert review and pilot testing. The scale comprises 6 items, rated on a 5-point Likert scale (1 = strongly disagree to 5 = strongly agree).
Change in Attitudes Toward Dementia | Baseline (Day 0, prior to intervention start) Immediate Post-Intervention (Day 0, following completion of the VR session, approximately 2 hours after Baseline assessment) Follow-up (Month 3, 12 weeks post-intervention, to assess retention effects)
  Attitudes toward dementia will be evaluated using the Dementia Attitude Scale (DAS), which has been adapted from the Attitudes Toward Dementia Scale (ATDS) and refined through expert review and pilot testing.
  The scale is made up of 10 items rated on a 5-point Likert scale, where 1 means "strongly disagree" and 5 means "strongly agree."

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan Normal University, Taipei, Taiwan